CLINICAL TRIAL: NCT02636374
Title: Guided Imagery: Reducing Stress and Improving Well-being in Pregnant Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-0105
Record Dates: First submitted 2015-12-01; First posted 2015-12-21 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Guided Imagery (Experimental): Participants listened to a pregnancy-specific guided imagery recording on four separate occasions during their pregnancies. Perceived stress was measured immediately pre and post each listening session using the Perceived Stress Measure-9 (PSM-9).
  Interventions: Behavioral: Guided Imagery

INTERVENTIONS:
Behavioral: Guided Imagery — A fifteen minute recording of gentle music together with soft talking to guide relaxation.

SUMMARY:
The purpose of this study is to examine the effects of a guided imagery intervention on perceived stress in pregnant adolescents.

DETAILED DESCRIPTION:
Pregnant adolescents attending a local alternative education program will be subjects of this study. Students will participate in four, 15 minute guided imagery sessions over about a 4-6 week period. They will complete a pregnancy specific stress questionnaire before beginning and after completion of the guided imagery protocol. The students will also complete a short 9-question stress measure before and after each of the individual guided imagery sessions.

The specific aims are:

1. to evaluate whether a guided imagery intervention reduces perceived stress in pregnant adolescents; and
2. to evaluate whether a guided imagery intervention enhances well-being in pregnant adolescents.

The hypotheses are that the intervention will reduce perceived stress and enhance well-being in these subjects. The purpose of this study is to assess whether employing a guided imagery intervention with pregnant teens and education will reduce perceived stress levels and improve well-being.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant students ages 13-21 enrolled in the alternative education program for parenting teens were eligible to participate

Exclusion Criteria:

* Participants were excluded from the study if they delivered their babies prior to completing four sessions of guided imagery intervention.

Ages: 13 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2012-11; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Change in Psychological Stress Measure-9 (PSM-9) score | 4 weeks
  Participants will complete the PSM-9 before and after listening to guided imagery sessions for each of the 4 weekly intervention sessions. The Psychological Stress Measure-9 (PSM-9) is a 9 item questionnaire measuring stress. The original form was published in Canada by Louise Lemyre, PHD and Rejean Tessier, PHD in 1988 and the 9 item was published in 2002. Each response rests on an 8 point likert scale. For general surveys of health and well-being in the workplace, an abridged 9-item version was developed to meet a variety of research needs and applications. The PSM-9 version is used at Hydro-Quebec and Renault (France) as well as in public service, hospitals, community services, and private practice. It has the same psychometric qualities of reliability, validity, and internal consistency (.89) and maintains the same heuristic value for statistics: normality of distribution and responsiveness (Lemyre, Chair, & Lalande-Markon, 2009).

CONTACTS AND LOCATIONS:
Overall Officials: Karla Ausderau, PhD, OTR/L, Principal Investigator — University of Wisconsin, Madison